CLINICAL TRIAL: NCT03741361
Title: The Impact of Anxiety or Depression on the Sedative Concentration of Propofol in Day-case Hysteroscopic Surgery: a Prospective Observational Study
Brief Title: The Impact of Anxiety or Depression on the Sedative Concentration of Propofol
Status: Completed | Type: Observational
Sponsor: Xuyu Zhang (Other)
Responsible Party: Sponsor-Investigator, Xuyu Zhang, Associate Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: SYSU 2018-11-02
Record Dates: First submitted 2018-11-11; First posted 2018-11-14 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Anxiety; Depression; Propofol; Anesthetics, Intravenous
Keywords: Female; Prospective Studies; Anesthetics, Intravenous; Propofol; Anxiety/*psychology; Depression/*psychology
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — An intravenous cannula was placed and 5 ml blood sample was drawn from each patient. The serum was separated and immediately stored at -80℃ for later analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anxiety and Depression: Female patients scheduled for hysteroscopic surgery under propofol-based intravenous anesthesia will be recruited in this prospective cohort study.
  Interventions: Other: anxiety and depression

INTERVENTIONS:
Other: anxiety and depression — Female patients who have a previous history of surgery or infertility, or a history of miscarriage or abortion are often susceptible to preoperative anxiety or depression. We will observe the effect of anxiety and depression on the dosage of propofol during induction.

SUMMARY:
120 consecutive female patients, 18-65 years old, American Society of Anesthesiologists (ASA) physical status I to II, scheduled for hysteroscopic surgery under propofol-based intravenous anesthesia will be recruited in this cohort study. The day before surgery, participants will be assessed the state of preoperative anxiety and depression. On the day of surgery, propofol will be administered by target controlled infusion (TCI) pump. During induction of anesthesia, the level of sedation will be evaluated. The induction dose of propofol, target effect-site concentration(Cet), plasma concentration(Cp) and effect-site concentration (Ce) of propofol will be recorded.

DETAILED DESCRIPTION:
120 consecutive female patients, 18-65 years old, American Society of Anesthesiologists ( ASA) physical status I to II, scheduled for hysteroscopic surgery under propofol-based intravenous anesthesia will be recruited in this prospective cohort study. The day before surgery, participants were asked to complete the modified HADS questionnaire in an isolated calm room, and the score was used to assess the patients' anxiety and depression level in the past 6 months. On the day of surgery, propofol (Fresenius Kabi Austria GmbH, Graz, Austria)was administrated by using an intravenous target controlled infusion (TCI) pump (Alaris PK, Basingstoke, UK) with Schnider kinetic model. The initial effect-site concentration (Ce) was set as 1.0 μg/ml. After the TCI system displayed that Cp and Ce were at equilibrium, the target concentration of propofol was increased by an increment of 0.5 μg/ml until the patients achieved the three desired levels of sedation.The Ce and dose of propofol and the consuming time were recorded.

ELIGIBILITY:
Inclusion Criteria:

* female
* American Society of Anesthesiologists（ASA） physical status I or II
* Body Mass Index(BMI) 18-25kg/m2
* scheduled for hysteroscopic surgery under propofol-based intravenous anesthesia.

Exclusion Criteria:

* suffering from psychiatric diseases.
* chronic use of anxiolytics, antidepressants, and sedative-hypnotics.
* any sedative premedication.
* a history of alcohol abuse.
* allergy to propofol.
* declining to participate and cooperate.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients, 18-65 years old, American Society of Anesthesiologists （ASA） physical status I or II, scheduled for hysteroscopic surgery under propofol-based intravenous anesthesia in the first affiliated hospital of Sun Yat-sen University in Guangzhou, China will be recruited in this cohort study.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Effect-site concentration (Ce) of propofol | Time of induction is less than 10 minutes.
  Effect-site concentration (Ce) of propofol on the TCI-system at the sedative level of OAA/S score of 3, OAA/S score of 1, and OAA/S core of 1 and NI<64 reached will be recorded.

SECONDARY OUTCOMES:
The induction dose of propofol | Time of induction is less than 10 minutes.
  The dose of propofol required at the sedative level of OAA/S score of 3, OAA/S score of 1, and OAA/S core of 1 and NI<64 reached will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Xuyu Zhang, M.D. and Ph.D, Principal Investigator — Department of Anesthesiology,The first affiliated hospital of Sun Yat-sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication.

REFERENCES:
- [Derived] Li RY, Lin M, Jiang HY, Wen SH, Shen JT, Huang WQ, Zhang XY. Impact of Anxiety or Depression Symptoms on Propofol Requirements for Sedation in Females: A Prospective Cohort Study. J Clin Pharmacol. 2020 Oct;60(10):1376-1384. doi: 10.1002/jcph.1631. Epub 2020 May 23. PMID 32445415